CLINICAL TRIAL: NCT00551616
Title: Safety and Efficacy of CDB-2914 in Comparison to Levonorgestrel for Emergency Contraception
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2914-004
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Contraception
MeSH Terms: interventions — ulipristal; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CDB-2914 (Experimental)
  Interventions: Drug: CDB-2914
- Levonorgestrel (Active Comparator)
  Interventions: Drug: Levonorgestrel

INTERVENTIONS:
Drug: CDB-2914 — Single dose
  Arms: CDB-2914
Drug: Levonorgestrel — Single dose
  Arms: Levonorgestrel

SUMMARY:
The purpose of this study is to assess the safety and efficacy of CDB-2914 in comparison to levonorgestrel for preventing pregnancy up to 5 days after unprotected sexual intercourse.

ELIGIBILITY:
Inclusion Criteria:

* women 16 or older in UK(except Northern Ireland) sites, 17 years or more in Northern Ireland (UK) and 18 years or more in Ireland and US
* present within 120 hours of unprotected intercourse
* regular menstrual cycles
* No current use of hormonal contraception
* Willing to not use hormonal methods of contraception until study completion
* At least one complete menstrual cycle (2 menses) post miscarriage, delivery or abortion
* For women who present more than 72 hours after intercourse, decline the insertion of an Intra Uterine Device for emergency contraception
* Able to provide informed consent
* Willing to abstain from further acts of unprotected intercourse until study completion

Exclusion Criteria:

* One or more acts of unprotected intercourse more than 120 hours
* current or recent use of hormonal methods of contraception
* currently pregnant or breastfeeding
* tubal ligation or current use of IUD
* Use of hormonal emergency contraception since last menstrual period
* Current use of IUD
* Tubal ligation
* Partner with a vasectomy
* Unsure about the date of the last menstrual period
* Severe asthma insufficiently controlled by oral glucocorticoid
* Hypersensitivity to the active substance levonorgestrel or any of the excipients of the drug products used in the study

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2221 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna F Glasier, MD, Principal Investigator — NHS Lothian Family Planning Service
Locations (33):
- United States (23):
  - Planned Parenthood Hollywood, Los Angeles, California
  - Planned Parenthood Santa Monica, Santa Monica, California
  - Planned Parenthood of the Rocky Mountains, Boulder, Colorado
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Planned Parenthood of the Rocky Mountains, Littleton, Colorado
  - Planned Parenthood of Greater Miami, Lake Worth, Florida
  - Planned Parenthood of Greater Miami, Miami, Florida
  - Planned Parenthood of Greater Miami, North Miami, Florida
  - Planned Parenthood of Greater Miami, Stuart, Florida
  - Planned Parenthood of Greater Miami, West Palm Beach, Florida
  - Planned Parenthood of Northeast Ohio Akron Health Center, Akron, Ohio
  - Planned Parenthood of Northeast Ohio Bedford Health Center, Bedford, Ohio
  - Planned Parenthood of Northeast Ohio East Cleveland Health Center, Cleveland, Ohio
  - Planned Parenthood of Northeast Ohio Old Brooklyn Health Center, Cleveland, Ohio
  - Planned Parenthood of Northeast Ohio Kent Health Center, Kent, Ohio
  - Planned Parenthood of Northeast Ohio Rocky River Health Center, Rocky River, Ohio
  - Planned Parenthood of Texas Capitol Region, Austin, Texas
  - Fannin Health Center, Houston, Texas
  - Planned Parenthood of Houston and Southeast Texas Research Department, Houston, Texas
  - Planned Parenthood Association of Utah, Ogden, Utah
  - Planned Parenthood Association of Utah, Orem, Utah
  - Planned Parenthood Association of Utah, Salt Lake City, Utah
  - Planned Parenthood Association of Utah, West Valley City, Utah
- Well Woman Centre, Dublin, Ireland
- United Kingdom (9):
  - NHS Grampian Sexual and Reproductive Health, Aberdeen
  - Brook Family Planning Clinic, Belfast
  - NHS Lothian Family Planning Service, Edinburgh
  - NHS Greater Glasgow & Clyde Family Planning Service, Glasgow
  - Liverpool PCT Family Planning Services, Liverpool
  - London Sexual and Reproductive Health, London
  - Manchester Primary Care Trust, Manchester
  - Nottingham Contraception & Sexual Health Service, Nottingham
  - Oxfordshire PCT Community Health, Oxford

REFERENCES:
- [Result] Glasier AF, Cameron ST, Fine PM, Logan SJ, Casale W, Van Horn J, Sogor L, Blithe DL, Scherrer B, Mathe H, Jaspart A, Ulmann A, Gainer E. Ulipristal acetate versus levonorgestrel for emergency contraception: a randomised non-inferiority trial and meta-analysis. Lancet. 2010 Feb 13;375(9714):555-62. doi: 10.1016/S0140-6736(10)60101-8. Epub 2010 Jan 29. PMID 20116841

RESULTS

PARTICIPANT FLOW:
Groups:
- CDB-2914: CDB-2914: Single dose (30 mg)
- Levonorgestrel: Levonorgestrel: Single dose (1.5 mg)
Period: Overall Study
Arm/Group | CDB-2914 | Levonorgestrel
Started | 1104 | 1117
Completed | 1056 | 1077
Not Completed | 48 | 40
Not completed — Lost to Follow-up | 48 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDB-2914 | Levonorgestrel | Total
Number analyzed (Participants) | 1104 | 1117 | 2221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 49 | 93
  Between 18 and 65 years | 1060 | 1068 | 2128
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (6.1) | 24.9 (6.5) | 24.7 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1104 | 1117 | 2221
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 804 | 809 | 1613
  Black | 210 | 207 | 417
  Asian | 13 | 21 | 34
  Other | 77 | 80 | 157
Time from unprotected sexual intercourse to emergency contraception (hours) [Count of Participants; unit: Participants]
  0-24h | 367 | 395 | 762
  25-48h | 388 | 378 | 766
  49-72h | 238 | 219 | 457
  73-96h | 72 | 86 | 158
  97-120h | 38 | 36 | 74
  >120h | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pregnancy
Description: The rate of pregnancy in women who received emergency contraception within 72 h of unprotected sexual intercourse.
Time Frame: Within 72 hours of unprotected Intercourse
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | CDB-2914 | Levonorgestrel
Number analyzed (Participants) | 1104 | 1117
Participants | 20 | 30

2. Secondary Outcome: Actual Pregnancy Rate Compared to Expected Pregnancy Rate
Description: Conditional probabilities of pregnancy from the time of unprotected sex intercourse to treatment were estimated for up to 120 hours using Spline Cubic Estimation (Stone & Koo, 1985) Pregnancy rate expected in the absence of emergency contraception is based on Trussell J, Rodriguez G, Ellertson C. New estimates of the effectiveness of the Yuzpe regimen of emergency contraception. Contraception. 1998;57(6):363-9.
Time Frame: Within 120 hours of unprotected Intercourse
Population: Efficacy evaluable population (women aged 35 years or younger who were enrolled for the first time in the study and whose pregnancy status after treatment was known)
Measure: Count of Participants; unit: Participants
Arm/Group | CDB-2914 | Levonorgestrel
Number analyzed (Participants) | 843 | 851
Participants
  Number of pregnancies observed | 15 | 22
  Number of expected pregnancies | 47 | 46
Statistical Analysis 1: Comparison: CDB-2914; Comparison of % of observed pregnancies vs % of expected pregnancies based on Trussell 1998; Test type: Other; p < 0.001, Chi-squared; % of observed pregnancies = 1.78, 95% CI 2-sided [1.04 to 2.98] — Expected pregnancy rate = 5.58%
Statistical Analysis 2: Comparison: Levonorgestrel; Comparison of % of observed pregnancies vs % of expected pregnancies based on Trussell 1998; Test type: Other; p < 0.001, Chi-squared; % of observed pregnancies = 2.59, 95% CI 2-sided [1.68 to 3.94] — Expected pregnancy rate = 5.43%

3. Secondary Outcome: Menstrual Bleeding Patterns
Description: Onset of next menses after emergency contraception compared to usual date.
Time Frame: within the menstrual cycle of the unprotected Intercourse
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: DAYS
Arm/Group | CDB-2914 | Levonorgestrel
Number analyzed (Participants) | 1104 | 1117
DAYS | 2.1 (8.2) | -1.2 (7.9)

ADVERSE EVENTS:
Time Frame: At the most 60 days after treatment.
Arm/Group | CDB-2914 | Levonorgestrel
All-Cause Mortality (participants affected / at risk) | 0/1104 | 0/1117
Serious Adverse Events (participants affected / at risk) | 3/1104 | 4/1117
Other Adverse Events (participants affected / at risk) | 596/1104 | 572/1117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDB-2914 (N=1104) | Levonorgestrel (N=1117)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Right contact lense related corneal ulcer (Eye disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Vomiting blood stained fluid (Gastrointestinal disorders) | 0 (0) | 1 (1)
Molar pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
ruptured ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDB-2914 (N=1104) | Levonorgestrel (N=1117)
Headache (Nervous system disorders) | 213 (213) | 211 (211)
Dysmenorrhoea (Reproductive system and breast disorders) | 142 (142) | 160 (160)
Nausea (Gastrointestinal disorders) | 141 (141) | 126 (126)
Abdominal pain (Gastrointestinal disorders) | 56 (56) | 75 (75)
Dizziness (Nervous system disorders) | 56 (56) | 55 (55)
Fatigue (General disorders) | 61 (61) | 44 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No